CLINICAL TRIAL: NCT02399033
Title: Xihuang Capsules Prevention of Recurrence in Patients With Hepatocellular Carcinoma After Hepatectomy: A Multicenter Randomized Controlled Trial
Brief Title: Xihuang Capsules Prevention of Recurrence in Patients With Hepatocellular Carcinoma After Hepatectomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shuqun Cheng (Other)
Responsible Party: Sponsor-Investigator, Shuqun Cheng, Xihuang Capsules prevention of recurrence in patients with hepatocellular carcinoma after hepatectomy: A multicenter randomized controlled trial., Eastern Hepatobiliary Surgery Hospital
Organization: Eastern Hepatobiliary Surgery Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SCheng
Record Dates: First submitted 2015-02-12; First posted 2015-03-26 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-02

CONDITIONS: Hepatocellular Carcinoma
Keywords: Xihuang Capsules; hepatocellular carcinoma; Recurrence; hepatectomy
MeSH Terms: conditions — Carcinoma, Hepatocellular; Recurrence | interventions — xihuang

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- the control group (No Intervention): Patients in Control group were not received Xihuang Capsules.
- Xihuang Capsules group (Experimental): Patients in Xihuang Capsules group were received Xihuang Capsules (2g, bid), Continuously taking to cancer recurrence or death.
  Interventions: Drug: Xihuang Capsules

INTERVENTIONS:
Drug: Xihuang Capsules — In two weeks after hepatectomy, Xihuang Capsules group received Xihuang Capsules (2 g, bid), Continuously taking to cancer recurrence or death.
  Other Names: Wangbang Pharmaceutical Xihuang Capsules
  Arms: Xihuang Capsules group

SUMMARY:
Study Objective: To evaluate the efficacy and safety of Xihuang Capsules prevention of recurrence in patients with hepatocellular carcinoma after hepatectomy.

Study Design: The study was A Multicenter, Randomized, Controlled, Open-Label, Parallel-Group Clinical Trial. Patients will be randomly assigned to Xihuang Capsules group or the control group by the proportion of 2: 1.

The total sample size: 1000 cases. Study Process: The study is divided into three phases: the screening phase, treatment phase, follow-up phase.To complete screening in two weeks, patients who fit the criteria were randomly assigned to Xihuang Capsules group or the control group.In two weeks after hepatectomy, Xihuang Capsules group received Xihuang Capsules (2g,bid), Continuously taking to cancer recurrence or death.Control group was not received Xihuang Capsules. In the first month to three years after treatment, Conducting visits for once every three months,to evaluate the efficacy and safety with hepatocellular carcinoma recurrence rate in the three years after hepatectomy as the primary outcome. When entering the follow-up phase, Keeping in touch with patients withdrew from the study for a clinic or telephone follow-up every three months.

From signing informed consent till the end of the study, inspecting the adverse events and concomitant medications for all subjects in each visit.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 20-70 years old;
2. Gender: male or female;
3. clinical or pathological diagnosis of hepatocellular carcinoma (HCC) in previously untreated patients;
4. The expected survival> 3 months;
5. Child-Pugh grade in A-level;
6. KPS score with 50-100 points;
7. In two weeks after hepatectomy for R0 resection surgery. Preoperative must meet the following criteria:

   * BCLC stage of 0-B;
   * conform to the indications of hepatectomy;
   * Viable tumor resection confirmed by two highly qualified surgical doctors;
   * No other surgical contraindications.
8. women in the reproductive period must be completely contraception in 28 days before treatment, during the treatment process and in 28 days after treatment;
9. Men must be completely contraception and prohibited donation and sperm donation during the treatment process and in 28 days after treatment;
10. All patients must be prohibited donation during the treatment process and in 28 days after treatment;
11. In addition to the subjects, prohibitting other people taking this product.
12. patients have a good understanding and could coordinate with investigators for the trial.
13. Patients enrolled in the trial should sign an informed consent form, to indicate understanding the purpose and procedure of the trial, and patients volunteering to participate in the trial.

Exclusion Criteria:

1. Because of suffering from any serious illness,laboratory abnormalities or mental abnormalities,the patient is unable to sign an informed consent form;
2. patients with medical abnormalities may result in that the trial could not be evaluated or have security risks;
3. persons who are unable to take oral drugs.
4. coagulation dysfunction;
5. HIV, syphilis-infected persons;
6. persons who have a serious heart, liver and renal failure;
7. persons who are known to allergic to the drug or any component of the drug;
8. persons who are received experimental therapy in 28 days before the first treatment;
9. persons who are received radiotherapy or other surgery(including of the other local surgery for cancer treatment,eg. TACE) in addition to hepatectomy in 14 days before the first treatment;
10. lactating or pregnant women;
11. patients in the reproductive period are unwilling or unable to contraception;
12. persons with poor medication compliance;
13. The researchers considered unsuitable selected patients.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2014-06; Primary Completion 2019-07 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Hepatocellular carcinoma recurrence rate in the three years after hepatectomy | in the three years after hepatectomy
  Diagnostic criteria for hepatocellular carcinoma recurrence: refer to Chinese Anti-Cancer Association Professional Committee of hepatocellular carcinoma developed diagnostic criteria for primary hepatocellular carcinoma belong to Guangzhou standard in 2001. Once new or suspected place nature lesions within liver were found by B-ultrasonography examination,we should do CT, MRI or PET-CT review, in order to confirm the diagnosis. If imaging is positive, diagnosing hepatocellular carcinoma(dominant) recurrence after treatment; if imaging is negative, but AFP values> 400μg/L or ongoing elevated AFP values, diagnosing hepatocellular carcinoma occult recurrence after treatment.

SECONDARY OUTCOMES:
Hepatocellular carcinoma recurrence rate in a year after hepatectomy | in a year after hepatectomy
Relapse free survival (RFS) | up to 5 years
  RFS is defined as from date of randomization until the date of first documented tumor recurrence or date of death from any cause, whichever came first.
Hepatocellular carcinoma survival rate in a year or three years after hepatectomy | in a year or three years after hepatectomy
Overall survival(OS) | up to 5 years
  OS is defined as from date of randomization until the date of documented death from any cause.
Improvement in quality of life in a year or three years after hepatectomy | in a year or three years after hepatectomy
  Using Karnofsky-Performance-Status score:
  Evaluation Methods: Comparison of symptom scores before and after the treatment.
  Markedly: increasing by more than 20 points after treatment compared to before treatment; Effective: increasing by more than 10 points after treatment compared to before treatment; Stable: increasing by less than 10 points or no change after treatment compared to before treatment; Invalid: decrease after treatment than before treatment.
number of participants with improvement of clinical symptoms, Such as flank pain, bloating, fatigue, anorexia and other syndromes of traditional Chinese Medicine. | participants will be followed for the duration of study, an expected average of 3 months.
  Evaluation index : according to clinical observations, TCM symptoms are divided into 4 levels: (0) no symptoms, (1) mild, (2) moderate, (3)severe, Recording treatment according to symptoms.
  Evaluation methods: comparison of symptom total integral before and after the treatment (before treatment / after treatment) Markedly: symptom disappeared, or symptom integral reduce ≥ 2/3; Effective: symptom alleviative, integral is reduced≥1/3，≤2/3; Invalid: symptom is not alleviated or reduced<1/3.
The incidence of adverse reaction. | up to 5 years
  Classification according to the Common Terminology Criteria Adverse Events Version 4.0(CTCAE v4.0).

CONTACTS AND LOCATIONS:
Overall Officials: Shuqun Cheng, Ph.D, Principal Investigator — Eastern Hepatobiliary Surgical Hospital
Locations (1):
- Eastern Hepatobiliary Surgical Hospital, Shanghai, Shanghai Municipality, China